CLINICAL TRIAL: NCT04827537
Title: Anti-protozoal Effect of Steroid Hormone 20-hydroxyecdysone
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan (Other Government)
Responsible Party: Principal Investigator, Svetlana Osipova, MD, PhD, DS, Dr., Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019121819
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Giardia Lamblia Infection
MeSH Terms: conditions — Giardiasis | interventions — Ecdysterone; Metronidazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 20-hydroxyecdysone group (Experimental): water sports athletes with Giardia infection will receive 20-hydroxyecdysone (100 mg (one pill) x two times a day orally), 10 consecutive days
  Interventions: Drug: 20-hydroxyecdysone Oral
- metronidazole group (Active Comparator): water sports athletes with Giardia infection will receive metronidazole, 500 mg (one pill) x two times a day orally, 10 consecutive days
  , and placebo preparations, respectively
  Interventions: Drug: Metronidazole Oral
- placebo group (Placebo Comparator): water sports athletes with Giardia infection will receive placebo preparation, 100 mg (one pill) x two times a day orally, 10 consecutive days
  Interventions: Drug: Placebo Oral

INTERVENTIONS:
Drug: 20-hydroxyecdysone Oral — 100 mg (one pill) x two times a day orally, 10 consecutive days
  Other Names: ecdysterone
  Arms: 20-hydroxyecdysone group
Drug: Metronidazole Oral — 500 mg (one pill) x two times a day orally, 10 consecutive days
  Other Names: Metronidazole
  Arms: metronidazole group
Drug: Placebo Oral — 100 mg (one pill) x two times a day orally, 10 consecutive days
  Other Names: shugar pills
  Arms: placebo group

SUMMARY:
20-hydroxyecdysone is an ecdysteroid hormone found in invertebrates and plants. 20-hydroxyecdysone exhibits a broad range of biological properties in various in vitro and in vivo models, including anabolic, antioxidant, anti-inflammatory, immunomodulatory, anti-obesity and antidiabetic activities, in addition to acting as neuroprotective and hepatoprotective agent. Ecdysteroids are widely used by athletes as dietary supplements to increase strength and muscle mass during resistance training, to reduce fatigue and to ease recovery. Mhashilkar AS et al. (2016) were revealed anti-parasitic activity of 20-hydroxyecdysone against the human filarial parasites. According to recent searches in academic databases and medical search engines (Google, www.google.com; PubMed, www.ncbi.nlm.nih.gov/pubmed; and Medline, www.medline.com), no studies have been conducted to assess the anti-protozoal activity of 20-hydroxyecdysone.

The aim of the study is to assess anti-protozoal activity of 20-hydroxyecdysone in water sports athletes with giardiasis.

DETAILED DESCRIPTION:
The randomized, double-blinded, placebo-controlled clinical study will be conducted by the Uzbek State University of Physical Education and Sport, Institute of the Chemistry of Plant Substances named acad. S. Yu. Yunusov and Republican Specialized Scientific and Practical Medical Center of Epidemiology, Microbiology, Infectious and Parasitic Diseases, Tashkent, Uzbekistan

Both informed and written consents will be obtained from the participants.

Study participants will be included about 200 athletes aged 18 to 27 years with giardiasis. All the participants will be residents of Uzbekistan.

Diagnosis of giardiasis will be based on the results of parasitological examination. Inclusion criteria:presence of giardia intestinalis in the stool samples of participant.

The exclusion criteria: chronic and acute infectious diseases, endocrine diseases, congenital diseases, allergic dermatitis, bronchial asthma, allergic rhinitis and/or conjunctivitis, other skin disorders, history of using vitamin D supplements within three months ago, or use of any medication influencing endocrine parameters.

Measurement of anthropometric indices Demographic data will be obtained in the survey included age, gender, and body mass index (BMI) calculated as weight (kg)/height2 (m2).

Blood Sample Collection and Storage Five milliliters of peripheral venous blood sample will be taken (after 8-12 hours of fasting) from each participant and will be collected into HumaTube Serum Gel - C/A for ELISA. Serum will be appropriately obtained and stored at -20°C maximum of 30 days. All blood samples will be collected before and after therapy.

200 water sports athletes with Giardia infection will be randomized from 1 to 3 groups to receive 20-hydroxyecdysone, metronidazole and placebo preparations, respectively

ELIGIBILITY:
Inclusion Criteria:

- a presence of giardia lamblia in stool samples of partisipants

Exclusion Criteria:

* chronic and acute infectious diseases,
* endocrine diseases, congenital diseases,
* allergic dermatitis,
* bronchial asthma,
* allergic rhinitis and/or conjunctivitis,
* other skin disorders,
* history of using vitamin D supplements within three months ago, or use of any medication influencing endocrine parameters.

Ages: 18 Years to 27 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Anti-protozoal effect of steroid hormone 20-hydroxyecdysone | up to 24 months
  Detection of Anti-protozoal effect of steroid hormone 20-hydroxyecdysone

CONTACTS AND LOCATIONS:
Overall Officials: Abdurakhim Toychiev, PhD, Study Chair — research institute of epidemiology, microbiology and infectious diseases
Locations (1):
- Research institute of epidemiology, microbiology and infectious diseases, Tashkent, Uchtepa, Uzbekistan